CLINICAL TRIAL: NCT00637104
Title: A European Multicenter, Randomized, Single Blind Study of the MAR-Tyn Cobalt Chromium TiN-Coated Balloon-Expandable Stent in the Treatment of Patients With de Novo Coronary Artery Lesions
Brief Title: European Multicenter, Randomized, Comparative Efficacy/Safety Study of the Mar-Tyn TiN-Coated Stent
Acronym: MARTIN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Biomedical Systems S.p.A. (Industry)
Responsible Party: prof. Aleardo Maresta, Head of Cardiology Department - S.Maria delle Croci Hospital, Ravenna (Italy)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBS/03-2007
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Artery Disease; Angioplasty, Transluminal, Percutaneous Coronary; Stents
Keywords: percutaneous transluminal coronary angioplasty; stents; restenosis; biocompatible materials; ceramics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - Mar-tyn (Experimental): It includes the implant of the Mar-tyn TiN coated stent
  Interventions: Device: Mar-Tyn TiN coated Co-Cr Numen stent implant
- B - Vision (Active Comparator): Includes all the patients treated with the Vision stent
  Interventions: Device: Vision Co-Cr stent implant

INTERVENTIONS:
Device: Mar-Tyn TiN coated Co-Cr Numen stent implant — Implant of the Mar-tyn TiN coated stent
  Other Names: Mar-Tyn; martin; TiN coated stent
  Arms: A - Mar-tyn
Device: Vision Co-Cr stent implant — Implant of the Vision stent
  Other Names: cobalt-chromium stent
  Arms: B - Vision

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the TiN-coated MAR-Tyn stent in maintaining minimum lumen diameter in de novo native coronary artery lesions as compared to an uncoated control cobalt-chromium balloon-expandable stent (Vision, Abbott Vascular). Both stents are mounted on a Rapid Exchange Stent Delivery System.

DETAILED DESCRIPTION:
Occlusive coronary artery disease is predominantly caused by coronary atherosclerosis, a pathologic vascular condition characterized by abnormal lipid and fibrous tissue accumulation in the vessel wall. This condition may be accompanied by degenerative changes and/or calcification leading to stenosis (narrowing) of the luminal channel. Percutaneous Transluminal Coronary Angioplasty (PTCA) is a well-accepted method of non-surgical myocardial revascularization for selected patients with symptomatic occlusive coronary artery disease.

Restenosis is the most important challenge limiting the long-term success of coronary angioplasty. Symptomatic restenosis usually occurs 6 months after an angioplasty procedure. The rates of restenosis reported in numerous clinical trials vary from 13% to 57%. This variability may be attributed in part to differences in the methods used to assess the occurrence of restenosis and in the criteria used to define restenosis. Regardless of the exact percentage, restenosis remains the Achilles heel of angioplasty. Numerous pharmaceutical approaches to limit restenosis have been tested, but none have been successful to date.

It was chosen to coat the stent with Titanium Nitrate (TiN), which is an inert, biocompatible material, that creates a thin physical barrier to diffusion of toxic metal atoms, TiN creates a very smooth surface that is impossible to obtain with a metal alloy. This coating was applied to the cobalt chromium platform, "Numen", made of the L605 Cobalt-20 Chromium-15 Tungsten-10 Nickel alloy. This alloy contains the lowest Nickel percentage of Cobalt Chromium alloys used for surgical implants. The strut thickness of the platform is reduced to the minimum of 65 microns for optimal hemodynamic performance and to permit an ultra low profile delivery system. The "Numen" design complies with the requirements of the "LMS -Less Mismatch Stent" theory applied where multiple 1 mm high zigzags form the stent pattern to align the segments at 45° with respect to blood flow when the stent is expanded to its nominal diameter. TiN coating is being used commercially for their hard-wearing and chemical inactive properties, particularly for surgical tools. TiN features chemical stability, great hardness, excellent wear properties, low electric impedance, biocompatibility, hemocompatibility and the possibility, through the application process, to exchange the orientation of the grains, the hardness, the wear characteristics and also the biocompatibility (a nanocrystalline structure produces a chemical surface more suitable for the endothelial cells). The produced coatings were very fine grained and dense with a porosity within the film structure of less than 10 nm in diameter. Furthermore, in an iliac artery stent model in normal rabbits, safety and efficacy in reduced restenosis of the TiN coated Numen™ stent was assessed.

The special TiN coating of the Mar-Tyn stents is very promising in reducing the lesions and the causes of intima neoplasia.

This study is a multicenter (up to 8 European centers), prospective, randomized single blind study. This study has a 2-arm design assessing the safety and effectiveness of the Tin-coated MAR-Tyn stent to an uncoated control cobalt-chromium balloon-expandable stent (Vision, Abbott Vascular), both mounted on a Rapid Exchange Stent Delivery System. A total of 160 patients will be entered in the study and will be randomized on a 1:1 basis. Patients who meet the eligibility criteria will be either randomized to Treatment A or Treatment B. The patient will not know which stent will be implanted while the physician will be unblinded . Patients will be followed at 30 days, 6, and 12 months post-procedure, with all patients undergoing repeat angiography at 6 months. All adverse events up to the 1 year follow-up period will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria:

1. The patient must be > 18 years of age;
2. Female of childbearing potential must have a negative pregnancy test within 7 days of enrollment and utilize reliable birth control for eight months after enrollment
3. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia;
4. Single treatment of de novo lesion in a major coronary artery in patients with single or multi-vessel disease; patients with multiple lesions can be included only if the other lesions do not require treatment;
5. Target vessel diameter at the lesion site is >2.50mm and <3.5mm in diameter (visual estimate);
6. Target lesion is >10mm and <22mm in length (visual estimate);
7. Target lesion stenosis is >50% and <100% (visual estimate);
8. At least TIMI II coronary flow;
9. Acceptable candidate for coronary artery bypass surgery (CABG);
10. Patient is willing to comply with the specified follow-up evaluation;
11. Patient must provide written informed consent prior to the procedure using a form that is approved by the local Ethics Committee.
12. Patient can be pre-treated with aspirin and clopidogrel or, alternatively, aspirin alone plus a loading dose of 300 mg of clopidogrel before procedure completion in case of urgent PCI

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
2. Has unstable angina classified as Braunwald III B or C and A I-II-III, or is having a peri infarction;
3. Unprotected left main coronary disease with >50% stenosis;
4. Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede runoff;
5. Have an ostial target lesion;
6. Have a target lesion in a venous graft;
7. Angiographic evidence of thrombus within target lesion;
8. Calcified lesion which cannot be successfully predilated;
9. Documented left ventricular ejection fraction <=25%;
10. Totally occluded vessel (TIMI 0 level);
11. Impaired renal function (creatinine > 3.0 mg/dl) at the time of treatment;
12. Pretreatment with devices other than balloon angioplasty;
13. Target lesion has excessive tortuousity or angulation (> 45°) which makes it unsuitable for stent delivery and deployment;
14. Target lesion involves bifurcation including a diseased side branch >=2 mm in diameter (either stenosis of both main vessel and major branch or stenosis of just major branch) that would require side branch stenting;
15. Prior stent within 5mm of target lesion;
16. Direct Stenting
17. Recipient of heart transplant;
18. Patient with a life expectancy less than 12 months;
19. Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix) and ticlopidine (Ticlid), heparin, cobalt, chromium, or contrast agent (that cannot be managed medically)
20. Recent (6 months) cerebrovascular accidents or intracranial hemorrhage
21. Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study;
22. Currently participating in an investigational drug or another device study;
23. Intervention of another lesion has occurred within 6 months before the index procedure;
24. In the investigator's opinion, the lesion is not suitable for stenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
in-stent minimum lumen diameter (MLD) | 6 months

SECONDARY OUTCOMES:
Composite of Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, thrombosis, or repeat target lesion revascularization | 30 days, 6 months, 12 months
Angiographic binary restenosis (>50% diameter stenosis) 6 months post-procedure. In-lesion minimum lumen diameter (MLD) at 6 months post-procedure. | 6 months
Target lesion revascularization (TLR) at 6 months post-procedure. Target vessel revascularization (TVR) at 6 months post-procedure. | 6 months
• Device success defined as achievement of a final residual diameter stenosis of <30% (by QCA), using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Balducelli, MD,FESC,FACC, Principal Investigator — Ospedale "S.Maria delle Croci" - Ravenna, Italy
Locations (7):
- Department of Internal Medicine III (Cardiology), University of Freiburg im Breisgau, Freiburg im Breisgau, Germany
- Italy (4):
  - Policlinico Universitario di Bari-Emodinamica Interventista, Bari, BA
  - Ospedale San Raffaele- Emodinamica e Cardiologia, Milan, MI
  - Ospedale di Ravenna, U.O. Cardiologia, Ravenna, Ra
  - Campus Biomedico, Cardiologia, Roma, Roma
- CARIM, Department of Cardiology, Maastricht, Netherlands
- Cardiocentro Ticino, Cardiologia, Lugano, Switzerland